CLINICAL TRIAL: NCT02087696
Title: Uncontrolled Study to Evaluate Efficacy of Tocilizumab in Patients With Moderate or Severe Rheumatoid Arthritis and Candidates With a Biological Monotherapy
Brief Title: Uncontrolled Study to Evaluate Efficacy of Tocilizumab in Patients With Moderate or Severe Rheumatoid Arthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Spanish Foundation of Rheumatology (Other)
Collaborators: Roche Farma, S.A (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FER-TOC-2013-01; 2013-004051-20 (EudraCT Number)
Record Dates: First submitted 2014-03-06; First posted 2014-03-14 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Arthritis, Rheumatoid
Keywords: Arthritis, Rheumatoid; methotrexate; intolerance; poor compliance; contraindication; Tocilizumab; monotherapy
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naive biological treatment (Other): Rheumatoid arthritis patients with intolerance or poor compliance or contraindication to methotrexate and who have not received previous biological treatment.
  Tocilizumab dose 8mg/kg administered every 4 weeks for 24 weeks
  Interventions: Drug: Tocilizumab
- Previous Biological treatment (Other): Rheumatoid arthritis patients with intolerance or poor compliance or contraindication to methotrexate and who have not received more than two previous biological treatments.
  Tocilizumab dose 8mg/kg administered every 4 weeks for 24 weeks
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab dose 8mg/kg administered every 4 weeks during 24 weeks.
  Other Names: RoActemra

SUMMARY:
The purpose of this project is to evaluate the efficacy of Tocilizumab (TCZ) given as monotherapy in patients with active rheumatoid arthritis (RA) according to EULAR response at 24 weeks after treatment initiation.

The study design is an intervention study, uncontrolled, multicenter, prospective, 32-weeks, two cohorts of patients with poor compliance or with any contraindication or intolerance to methotrexate.

One cohort naive to previous biological therapy and the other one treated previously with a biological treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ability and willing to provide written informed consent and comply with the requirements of the study protocol.
* Patients with active moderate or severe rheumatoid arthritis, according to 1987 ACR criteria, diagnosed at least 6 months before inclusion.
* 18 years old or older
* DAS28 index greater than 3.2 at baseline.
* If patients are receiving corticosteroid the dose will have to be ≤ 10 mg of prednisone (or equivalent) and the patient must have been stable for at least one month previous to initiating treatment with Tocilizumab (day 1). Patients may have been treated with nonsteroidal antiinflammatory drug (NSAIDs) at stable doses during the previous month to inclusion.
* Patients receiving outpatient treatment.
* Women of childbearing potential and men with childbearing potential partners may only participate in the study if they use reliable contraception (eg barrier methods [the patient or her partner], oral or patch contraceptives, spermicide and barrier method or intrauterine device) during the study period and at least 3 months after receiving the last dose of Tocilizumab.
* In women of childbearing potential the pregnancy test must be negative at the screening visit and at baseline.
* Patients on methotrexate monotherapy or combined treatment with a biological agent, or patients on biological treatment monotherapy, who show or have ever shown intolerance or poor compliance or safety issues with methotrexate.
* Patients judge to be candidates to biological monotherapy by the researcher, without excluding previous use of other disease-modifying antirheumatic drug (DMARDs) different to methotrexate.

Exclusion Criteria:

* Patients with no peripheral venous access.
* Patients with previous failure to more than two biological treatments.
* Previous treatment with Tocilizumab at any time before the baseline visit.
* Treatment with any other agent on research during the four weeks previous to the screening visit (or equivalent period to its five half-lives) Considering the longest period.
* Previous treatment with cell depletion therapies, including experimental treatments or approved agents, as for examples: CAMPATH, antiCD4, antiCD5, antiCD3, antiCD19 and antiCD20).
* Treatment with intravenous gammaglobulin or plasmapheresis in the 6 months previous to the baseline visit.
* Intra-articular or parenteral corticosteroids within 4 weeks previous to the baseline visit.
* Immunization with a live / attenuated vaccine in the previous 4 weeks to the baseline visit.
* Previous treatment with alkylating agents such as chlorambucil, or full lymphoid irradiation.
* History of severe allergic or anaphylactic reactions to human, humanized or murine, monoclonal antibodies.
* Evidence of serious uncontrolled concomitant disease: cardiovascular, nervous system, lung (including chronic obstructive pulmonary disease), renal, hepatic, endocrine (including uncontrolled diabetes mellitus) or gastrointestinal.
* History of diverticulitis, diverticulosis requiring treatment with antibiotics, or chronic lower gastrointestinal ulcer disease, Crohn's disease, ulcerative colitis or any other lower gastrointestinal symptomatic conditions that could predispose to perforations.
* Known active Infections, or a history of known recurring infections: Mycobacterial, fungal, viral or bacterial type (included, but not limited to, tuberculosis, atypical mycobacterial disease, hepatitis B and C, herpes zoster, but excluding nail bed fungal infections).
* Any major episode of infection that required hospitalization or treatment with intravenous antibiotics within 4 weeks previous to the screening visit or oral antibiotics within 2 weeks previous to the screening visit.
* Active tuberculosis requiring treatment in the past year. Latent tuberculosis screening will be perform on all patients according to Spanish Society of Rheumatology/Spanish Agency for Medicines and Health Products (SER/AEMPS) guidelines of the. Patients treated for tuberculosis without recurrence in the past 3 years will not be excluded.
* Ongoing liver disease as determined by the principal investigator.
* Evidence of active malignancy, malignancies diagnosed in the previous 10 years (including solid and hematologic tumors, except basal cell carcinoma and squamous cell skin or removed and cured in situ cervix carcinoma), or breast cancer diagnosed in the previous 20 years.
* Pregnant or breastfeeding women.
* Patients with reproductive potential who are unwilling to use effective contraception.
* History of alcoholism, drug abuse or addiction in the previous year to the screening visit.
* Neuropathies or other painful conditions that may interfere with pain assessment.
* Serum creatinine >1,4 mg/dl (124 mol/l) in women and >1.6 mg/dl (141 mol/l) in men.
* Alanine aminotransferase or aspartate aminotransferase > 1.5 times the upper limit of normal.
* Total bilirubin greater than the upper limit of normal.
* Platelet count minor than 100 x 10^9/l (100.000/mm3).
* Hemoglobin minor than 85 g/L (<8,5 g/dL, 5,3 mmol/L).
* Leukocytes minor than 3,0 x 10^9/L (3000/mm3).
* Neutrophils, absolute value minor than 2,0 x 10^9/L (2000/mm3).
* Lymphocytes, absolute value minor than 0,5 x 10^9 /L (500/mm3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-12 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients achieving good or moderate European League Against Rheumatism (EULAR) response. | At 24 weeks of treatment.
  To evaluate the efficacy of Tocilizumab monotherapy administered in patients with active rheumatoid arthritis, in terms of percentage of patients achieving good or moderate European League Against Rheumatism (EULAR) response. To be classified as a good response, patients must have a clinically significant change (> 1.2) in DAS28 index as well as achieving low disease activity. Moderate answer assumes DAS28 index decreases between 0.6 and 1,2, long as it reaches low or moderate disease activity (DAS28 ≤ 5.1), or clinically significant (> 1.2) in the DAS28 in patients with a moderate or high activity (DAS28> 3.2) is achieved.

SECONDARY OUTCOMES:
Changes in the mean of DAS28 index. | Between baseline and week 24.
  To evaluate the efficacy of Tocilizumab monotherapy administered in patients with active rheumatoid arthritis, in terms of Disease Activity Score 28 (DAS28) change by the response EULAR criteria.
Changes in the mean of Simplex Disease Activity Index (SDAI), Clinical Disease Activity Index (CDAI). | At 24 weeks of treatment.
  To evaluate the activity of rheumatoid arthritis by the Simplex Disease Activity Index (SDAI), Clinical Disease Activity Index (CDAI) using the mean change in these index.
Percentage of patients complying American College of Rheumatology (ACR) criteria (ACR20, ACR50 and ACR70). | At 24 weeks of treatment
  To evaluate the efficacy by the American College of Rheumatology (ACR) criteria.
Changes in the mean of DAS28 index into several subgroups. | between baseline and week 24
  To evaluate the efficacy in patients with active rheumatoid arthritis treated with Tocilizumab monotherapy by the change in DAS28 index between baseline and week 24 in the following subgroups:
  Baseline DAS28: greater than 3.2 and less than 5.1 Baseline DAS28: greater than or equal to 5.1 Cohort A: Patients who have never been treated with biological therapy. Cohort B: Patients who have been previously treated with biological therapy.
Percentage of patients with a DAS28 index less than or equal to 3.2 | At week 24 of treatment.
Number of non-serious, serious or unexpected adverse events. | At the end of study (32 weeks).
  To evaluate the safety of Tocilizumab monotherapy during the study period.
Changes in the mean of Health-Related Quality of Life (HRQOL) index into several subgroups. | between baseline and week 24.
  To evaluate the Health-Related Quality of Life (HRQOL) of patients with rheumatoid arthritis treated with Tocilizumab monotherapy in the following subgroups:
  Baseline DAS28: greater than 3.2 and less than 5.1 Baseline DAS28: greater than or equal to 5.1 Cohort A: Patients who have never been treated with biological therapy. Cohort B: Patients who have been previously treated with biological therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Marsal Barril, MD; PhD, Principal Investigator — Hospital Vall d'Hebron
Locations (20):
- Spain (20):
  - Hospital Universitario Araba (Sede Txagorritxu), Vitoria-Gasteiz, Alava
  - Hospital del la Agencia Valenciana de Salud Vega Baja, Orihuela, Alicante
  - Hospital Can Misses, Ibiza Town, Balearic Islands
  - Hospital Universitari Son Espases, Mallorca, Balearic Islands
  - Hospital Universitari Vall d´Hebron, Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Puerta del Mar, Cadiz, Cádiz
  - Hospital Universitario Reina Sofía, Córdoba, Córdoba
  - Hospital San Cecilio, Granada, Granada
  - Hospital Universitario de Guadalajara, Guadalajara, Guadalajara
  - Complejo hospitalario Universitario de A Coruña, A Coruña, La Coruña
  - Complejo Asistencial Universitario de León, León, León
  - Hospital Universitario de La Princesa, Madrid, Madrid
  - Hospital Civil, Málaga, Málaga
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz de Tenerife
  - Hospital de Sagunto, Sagunto, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia, Valencia
  - Hospital Galdakao-Usansolo, Galdakao, Vizcaya

REFERENCES:
- [Background] Carmona L, Villaverde V, Hernandez-Garcia C, Ballina J, Gabriel R, Laffon A; EPISER Study Group. The prevalence of rheumatoid arthritis in the general population of Spain. Rheumatology (Oxford). 2002 Jan;41(1):88-95. doi: 10.1093/rheumatology/41.1.88. PMID 11792885
- [Background] Lajas C, Abasolo L, Bellajdel B, Hernandez-Garcia C, Carmona L, Vargas E, Lazaro P, Jover JA. Costs and predictors of costs in rheumatoid arthritis: a prevalence-based study. Arthritis Rheum. 2003 Feb 15;49(1):64-70. doi: 10.1002/art.10905. PMID 12579595
- [Background] Carmona L, Ballina J, Gabriel R, Laffon A; EPISER Study Group. The burden of musculoskeletal diseases in the general population of Spain: results from a national survey. Ann Rheum Dis. 2001 Nov;60(11):1040-5. doi: 10.1136/ard.60.11.1040. PMID 11602475
- [Background] Smolen JS, Landewe R, Breedveld FC, Dougados M, Emery P, Gaujoux-Viala C, Gorter S, Knevel R, Nam J, Schoels M, Aletaha D, Buch M, Gossec L, Huizinga T, Bijlsma JW, Burmester G, Combe B, Cutolo M, Gabay C, Gomez-Reino J, Kouloumas M, Kvien TK, Martin-Mola E, McInnes I, Pavelka K, van Riel P, Scholte M, Scott DL, Sokka T, Valesini G, van Vollenhoven R, Winthrop KL, Wong J, Zink A, van der Heijde D. EULAR recommendations for the management of rheumatoid arthritis with synthetic and biological disease-modifying antirheumatic drugs. Ann Rheum Dis. 2010 Jun;69(6):964-75. doi: 10.1136/ard.2009.126532. Epub 2010 May 5. PMID 20444750
- [Background] Knevel R, Schoels M, Huizinga TW, Aletaha D, Burmester GR, Combe B, Landewe RB, Smolen JS, Sokka T, van der Heijde DM. Current evidence for a strategic approach to the management of rheumatoid arthritis with disease-modifying antirheumatic drugs: a systematic literature review informing the EULAR recommendations for the management of rheumatoid arthritis. Ann Rheum Dis. 2010 Jun;69(6):987-94. doi: 10.1136/ard.2009.126748. Epub 2010 May 6. PMID 20448280
- [Background] Eberhardt K, Fex E. Clinical course and remission rate in patients with early rheumatoid arthritis: relationship to outcome after 5 years. Br J Rheumatol. 1998 Dec;37(12):1324-9. doi: 10.1093/rheumatology/37.12.1324. PMID 9973158
- [Background] Goekoop-Ruiterman YP, de Vries-Bouwstra JK, Allaart CF, van Zeben D, Kerstens PJ, Hazes JM, Zwinderman AH, Ronday HK, Han KH, Westedt ML, Gerards AH, van Groenendael JH, Lems WF, van Krugten MV, Breedveld FC, Dijkmans BA. Clinical and radiographic outcomes of four different treatment strategies in patients with early rheumatoid arthritis (the BeSt study): a randomized, controlled trial. Arthritis Rheum. 2005 Nov;52(11):3381-90. doi: 10.1002/art.21405. PMID 16258899
- [Background] Aletaha D, Stamm T, Kapral T, Eberl G, Grisar J, Machold KP, Smolen JS. Survival and effectiveness of leflunomide compared with methotrexate and sulfasalazine in rheumatoid arthritis: a matched observational study. Ann Rheum Dis. 2003 Oct;62(10):944-51. doi: 10.1136/ard.62.10.944. PMID 12972472
- [Background] De La Mata J, Blanco FJ, Gomez-Reino JJ. Survival analysis of disease modifying antirheumatic drugs in Spanish rheumatoid arthritis patients. Ann Rheum Dis. 1995 Nov;54(11):881-5. doi: 10.1136/ard.54.11.881. PMID 7492236
- [Background] Galindo-Rodriguez G, Avina-Zubieta JA, Russell AS, Suarez-Almazor ME. Disappointing longterm results with disease modifying antirheumatic drugs. A practice based study. J Rheumatol. 1999 Nov;26(11):2337-43. PMID 10555887
- [Background] Grove ML, Hassell AB, Hay EM, Shadforth MF. Adverse reactions to disease-modifying anti-rheumatic drugs in clinical practice. QJM. 2001 Jun;94(6):309-19. doi: 10.1093/qjmed/94.6.309. PMID 11391029
- [Background] Fitzpatrick R, Scott DG, Keary I. Cost-minimisation analysis of subcutaneous methotrexate versus biologic therapy for the treatment of patients with rheumatoid arthritis who have had an insufficient response or intolerance to oral methotrexate. Clin Rheumatol. 2013 Nov;32(11):1605-12. doi: 10.1007/s10067-013-2318-z. Epub 2013 Jul 9. PMID 23835658
- [Background] DiMatteo MR. Variations in patients' adherence to medical recommendations: a quantitative review of 50 years of research. Med Care. 2004 Mar;42(3):200-9. doi: 10.1097/01.mlr.0000114908.90348.f9. PMID 15076819
- [Background] van den Bemt BJ, Zwikker HE, van den Ende CH. Medication adherence in patients with rheumatoid arthritis: a critical appraisal of the existing literature. Expert Rev Clin Immunol. 2012 May;8(4):337-51. doi: 10.1586/eci.12.23. PMID 22607180
- [Background] Waimann CA, Marengo MF, de Achaval S, Cox VL, Garcia-Gonzalez A, Reveille JD, Richardson MN, Suarez-Almazor ME. Electronic monitoring of oral therapies in ethnically diverse and economically disadvantaged patients with rheumatoid arthritis: consequences of low adherence. Arthritis Rheum. 2013 Jun;65(6):1421-9. doi: 10.1002/art.37917. PMID 23728826
- [Background] Morand EF, McCloud PI, Littlejohn GO. Life table analysis of 879 treatment episodes with slow acting antirheumatic drugs in community rheumatology practice. J Rheumatol. 1992 May;19(5):704-8. PMID 1613698
- [Background] Askling J, Fored CM, Brandt L, Baecklund E, Bertilsson L, Feltelius N, Coster L, Geborek P, Jacobsson LT, Lindblad S, Lysholm J, Rantapaa-Dahlqvist S, Saxne T, van Vollenhoven RF, Klareskog L. Time-dependent increase in risk of hospitalisation with infection among Swedish RA patients treated with TNF antagonists. Ann Rheum Dis. 2007 Oct;66(10):1339-44. doi: 10.1136/ard.2006.062760. Epub 2007 Jan 29. PMID 17261532
- [Background] Heiberg MS, Koldingsnes W, Mikkelsen K, Rodevand E, Kaufmann C, Mowinckel P, Kvien TK. The comparative one-year performance of anti-tumor necrosis factor alpha drugs in patients with rheumatoid arthritis, psoriatic arthritis, and ankylosing spondylitis: results from a longitudinal, observational, multicenter study. Arthritis Rheum. 2008 Feb 15;59(2):234-40. doi: 10.1002/art.23333. PMID 18240258
- [Background] Lee SJ, Chang H, Yazici Y, Greenberg JD, Kremer JM, Kavanaugh A. Utilization trends of tumor necrosis factor inhibitors among patients with rheumatoid arthritis in a United States observational cohort study. J Rheumatol. 2009 Aug;36(8):1611-7. doi: 10.3899/jrheum.080889. Epub 2009 Apr 15. PMID 19369454
- [Background] Listing J, Strangfeld A, Rau R, Kekow J, Gromnica-Ihle E, Klopsch T, Demary W, Burmester GR, Zink A. Clinical and functional remission: even though biologics are superior to conventional DMARDs overall success rates remain low--results from RABBIT, the German biologics register. Arthritis Res Ther. 2006;8(3):R66. doi: 10.1186/ar1933. Epub 2006 Apr 5. PMID 16600016
- [Background] Mariette X, Gottenberg JE, Ravaud P, Combe B. Registries in rheumatoid arthritis and autoimmune diseases: data from the French registries. Rheumatology (Oxford). 2011 Jan;50(1):222-9. doi: 10.1093/rheumatology/keq368. PMID 21148156
- [Background] Sarzi-Puttini P, Antivalle M, Marchesoni A, Favalli EG, Gorla R, Filippini M, Caporali R, Bobbio-Pallavicini F, Montecucco C, Atzeni F. Efficacy and safety of anti-TNF agents in the Lombardy rheumatoid arthritis network (LORHEN). Reumatismo. 2008 Oct-Dec;60(4):290-5. doi: 10.4081/reumatismo.2008.290. PMID 19132154
- [Background] Soliman MM, Ashcroft DM, Watson KD, Lunt M, Symmons DP, Hyrich KL; British Society for Rheumatology Biologics Register. Impact of concomitant use of DMARDs on the persistence with anti-TNF therapies in patients with rheumatoid arthritis: results from the British Society for Rheumatology Biologics Register. Ann Rheum Dis. 2011 Apr;70(4):583-9. doi: 10.1136/ard.2010.139774. Epub 2011 Feb 17. PMID 21330639
- [Background] Yazici Y, Shi N, John A. Utilization of biologic agents in rheumatoid arthritis in the United States: analysis of prescribing patterns in 16,752 newly diagnosed patients and patients new to biologic therapy. Bull NYU Hosp Jt Dis. 2008;66(2):77-85. PMID 18537774
- [Background] Dougados M, Kissel K, Sheeran T, Tak PP, Conaghan PG, Mola EM, Schett G, Amital H, Navarro-Sarabia F, Hou A, Bernasconi C, Huizinga TW. Adding tocilizumab or switching to tocilizumab monotherapy in methotrexate inadequate responders: 24-week symptomatic and structural results of a 2-year randomised controlled strategy trial in rheumatoid arthritis (ACT-RAY). Ann Rheum Dis. 2013 Jan;72(1):43-50. doi: 10.1136/annrheumdis-2011-201282. Epub 2012 May 5. PMID 22562983
- [Background] Jones G, Sebba A, Gu J, Lowenstein MB, Calvo A, Gomez-Reino JJ, Siri DA, Tomsic M, Alecock E, Woodworth T, Genovese MC. Comparison of tocilizumab monotherapy versus methotrexate monotherapy in patients with moderate to severe rheumatoid arthritis: the AMBITION study. Ann Rheum Dis. 2010 Jan;69(1):88-96. doi: 10.1136/ard.2008.105197. PMID 19297346
- [Background] Bykerk VP, Ostor AJ, Alvaro-Gracia J, Pavelka K, Ivorra JA, Graninger W, Bensen W, Nurmohamed MT, Krause A, Bernasconi C, Stancati A, Sibilia J. Tocilizumab in patients with active rheumatoid arthritis and inadequate responses to DMARDs and/or TNF inhibitors: a large, open-label study close to clinical practice. Ann Rheum Dis. 2012 Dec;71(12):1950-4. doi: 10.1136/annrheumdis-2011-201087. Epub 2012 May 21. PMID 22615456
- [Background] Emery P, Keystone E, Tony HP, Cantagrel A, van Vollenhoven R, Sanchez A, Alecock E, Lee J, Kremer J. IL-6 receptor inhibition with tocilizumab improves treatment outcomes in patients with rheumatoid arthritis refractory to anti-tumour necrosis factor biologicals: results from a 24-week multicentre randomised placebo-controlled trial. Ann Rheum Dis. 2008 Nov;67(11):1516-23. doi: 10.1136/ard.2008.092932. Epub 2008 Jul 14. PMID 18625622
- [Background] Lingjaerde O, Ahlfors UG, Bech P, Dencker SJ, Elgen K. The UKU side effect rating scale. A new comprehensive rating scale for psychotropic drugs and a cross-sectional study of side effects in neuroleptic-treated patients. Acta Psychiatr Scand Suppl. 1987;334:1-100. doi: 10.1111/j.1600-0447.1987.tb10566.x. No abstract available. PMID 2887090
- [Background] Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Med Care. 1986 Jan;24(1):67-74. doi: 10.1097/00005650-198601000-00007. PMID 3945130
- [Background] Carmona L, Gomez-Reino JJ, Rodriguez-Valverde V, Montero D, Pascual-Gomez E, Mola EM, Carreno L, Figueroa M; BIOBADASER Group. Effectiveness of recommendations to prevent reactivation of latent tuberculosis infection in patients treated with tumor necrosis factor antagonists. Arthritis Rheum. 2005 Jun;52(6):1766-72. doi: 10.1002/art.21043. PMID 15934089